CLINICAL TRIAL: NCT00851253
Title: The Feasibility and Outcome of Cyberknife® Stereotactic Radiosurgical Boost and Salvage Therapy for Head and Neck Cancer
Brief Title: Stereotactic Radiosurgery in Treating Patients With Locally Advanced or Recurrent Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Minh Tam Truong, BMC Attending Physician, Boston Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-26649; W912SQ7058N601 (Other Grant/Funding Number: Dept of Defense)
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Head and Neck Cancer
Keywords: recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; stage II salivary gland cancer; stage III salivary gland cancer; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; stage IV salivary gland cancer; stage IV lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV basal cell carcinoma of the lip
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (CK SRS boost therapy) (Experimental): Radiation: CyberKnife Stereotactic Radiosurgery boost (2 fractionated doses) beginning 4-8 weeks after completion of standard therapy.
  Interventions: Radiation: stereotactic radiosurgery
- Group 2 (CK SRS salvage therapy) (Experimental): Radiation : CyberKnife® stereotactic radiosurgery salvage therapy (5 fractions) 3 times weekly.
  Interventions: Radiation: stereotactic radiosurgery

INTERVENTIONS:
Radiation: stereotactic radiosurgery — Given in 2 fractionated doses or 5 fractionated doses
  Other Names: CyberKnife

SUMMARY:
RATIONALE: Stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects of stereotactic radiosurgery in treating patients with locally advanced or recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the feasibility and tolerability of CyberKnife® stereotactic radiosurgery as boost therapy after standard chemoradiotherapy in patients with locally advanced head and neck cancer.
* To determine the feasibility and tolerability of CyberKnife® stereotactic radiosurgery as salvage therapy in patients with locally recurrent head and neck cancer.

OUTLINE: Patients are assigned to 1 of 2 treatment groups according to disease status after prior standard therapy. Patients with residual disease after standard therapy are assigned to group 1. Patients with recurrent disease ≥ 6 months after standard therapy are assigned to group 2.

All patients undergo placement of 3-6 gold fiducial markers within 1-2 weeks of beginning CyberKnife® stereotactic radiosurgery (SRS) treatment.

* Group 1 (CyberKnife® SRS boost therapy): Patients undergo CyberKnife® SRS boost therapy (2 fractionated doses) beginning 4-8 weeks after completion of standard therapy.
* Group 2 (CyberKnife® SRS salvage therapy): Patients undergo CyberKnife® SRS salvage therapy (5 fractions) 3 times weekly.

After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Biopsy-confirmed* invasive head and neck cancer, including the following primary sites:

  * Nasopharynx
  * Oropharynx
  * Paranasal sinus
  * Oral cavity
  * Orbit
  * Salivary gland NOTE: *Biopsy must be performed prior to initiation of external beam radiotherapy (EBRT)
* Stage T2-4 tumor at the time of diagnosis

  * Primary tumor ≤ 5 cm in diameter at the time of CyberKnife® stereotactic radiosurgery (SRS)
* Meets one of the following criteria:

  * Eligible for CyberKnife® SRS as boost therapy, as defined by one of the following criteria:

    * Planning to undergo definitive EBRT, with or without chemotherapy, with curative intent for primary head and neck cancer
    * Biopsy-confirmed locally persistent disease < 3 months after completion of definitive EBRT
  * Eligible for CyberKnife® SRS as salvage therapy*, as defined by one of the following criteria:

    * Biopsy-confirmed locally recurrent disease occurring ≥ 6 months after the completion of radiotherapy; achieved a complete response to initial therapy by imaging or clinical examination; had > 50% of the tumor volume in the prior irradiated volume; and received > 45 Gy of radiotherapy
    * Biopsy-confirmed locally recurrent disease occurring between 6 weeks and 6 months after the completion of radiotherapy; achieved a complete response to initial therapy by imaging or clinical examination; had < 50% of the tumor volume in the prior irradiated volume; and received > 45 Gy of radiotherapy NOTE: *Not a candidate for salvage surgery or brachytherapy
* Anticipated total dose of radiotherapy to the spinal cord ≤ 50 Gy (including prior dose)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to achieve normal tissue tolerance to critical structures with the CyberKnife® planning system
* Able to undergo CT simulation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Exclusion Criteria:

* No laryngeal or hypopharyngeal cancer
* No evidence of distant metastases
* No prior brachytherapy
* No prior CyberKnife® SRS boost or salvage therapy
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No active connective tissue disorders (e.g., lupus or scleroderma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minh T. Truong, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from within the investigators clinic practice between February 2009 and August 2013
Pre-assignment Details: One subject that was enrolled onto the Boost Arm was withdrawn prior to undergoing cyberknife therapy due to disease progression.
Period: Overall Study
Arm/Group | Group 1 (CK SRS Boost Therapy) | Group 2 (CK SRS Salvage Therapy)
Started | 2 | 10
Completed | 1 | 10
Not Completed | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (CK SRS Boost Therapy) | Group 2 (CK SRS Salvage Therapy) | Total
Number analyzed (Participants) | 2 | 10 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 5
  >=65 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 0 | 6 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Local Control
Description: Median time to local failure based on regional or distant metastatic disease
Time Frame: 1 year
Population: Boost subjects were not evaluable.
Measure: Median (Standard Deviation); unit: number of months to local failure
Arm/Group | Group 1 (CK SRS Boost Therapy) | Group 2 (CK SRS Salvage Therapy)
Number analyzed (Participants) | 0 | 10
number of months to local failure |  | 4.6 (1.6)

2. Secondary Outcome: Rates of Adverse Events Associated With Treatment
Description: Number of patients with serious adverse events possibly related, probably related or definitely related to the study treatment
Time Frame: 1 year
Population: One subject in the Boost Arm was withdrawn prior to Cyberknife therapy due to disease progression and was therefore not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (CK SRS Boost Therapy) | Group 2 (CK SRS Salvage Therapy)
Number analyzed (Participants) | 1 | 10
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group 1 (CK SRS Boost Therapy) | Group 2 (CK SRS Salvage Therapy)
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/1 | 9/10
Other Adverse Events (participants affected / at risk) | 1/1 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (CK SRS Boost Therapy) (N=1) | Group 2 (CK SRS Salvage Therapy) (N=10)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
pain (General disorders) | 1 (1) | 2 (2)
dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1)
dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ulceration (General disorders) | 0 (0) | 1 (1)
hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hemoglobinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
osteomyelitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (CK SRS Boost Therapy) (N=1) | Group 2 (CK SRS Salvage Therapy) (N=10)
pain (General disorders) | 0 (0) | 4 (4)
anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 2 (3)
dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
edema - head and neck (General disorders) | 1 (1) | 3 (3)
dizziness (Nervous system disorders) | 1 (1) | 1 (1)
fatigue (General disorders) | 1 (1) | 2 (2)
gait disturbance (Gastrointestinal disorders) | 1 (1) | 0 (0)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
lypmphatics disorder - other (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — moderate secretions from tracheotomy
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
taste alteration (Gastrointestinal disorders) | 0 (0) | 2 (2)
neurology - other (Nervous system disorders) | 0 (0) | 1 (2) — headaches 6/10 at worst controlled with pain medication
dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
weight loss (Investigations) | 0 (0) | 3 (3)
voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
mucositis (Gastrointestinal disorders) | 0 (0) | 2 (2)
dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No